CLINICAL TRIAL: NCT03837847
Title: Mechanistic Effects of Health Coaching to Reduce COPD Hospitalizations
Brief Title: Mechanistic Effects of Health Coaching to Reduce Chronic Obstructive Pulmonary Disease (COPD) Hospitalizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-000780; 1K24HL138150-01A1 (NIH)
Record Dates: First submitted 2019-01-21; First posted 2019-02-12 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: COPD; Emphysema
Keywords: Health coaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Intervention Model Description: Randomized Control wait design
Masking Description: It is not possible to blind the participants or the study team as subjects will know if they are receiving a health coaching call.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): Participants in this group will receive health coaching calls
  Interventions: Behavioral: Health Coaching Calls
- Control group (Active Comparator): Participants in this group will receive 6 educational guides
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Health Coaching Calls — Participants in this group will receive 12 weekly health coaching calls
  Arms: Health Coaching
Behavioral: Control — Participants in this group will receive 6 educational guides
  Arms: Control group

SUMMARY:
The researchers are trying to explore the benefit of Health Coaching on patients with severe symptoms of COPD.

ELIGIBILITY:
Inclusion Criteria: Men and women 40 years or older with a clinical diagnosis of COPD with shortness of breath.

Exclusion: terminal illness, inability to communicate by phone

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Participants in this group received 6 educational guides and 6 calls
  Control: Participants in this group received 6 educational guides and 6 calls to remind them to read the educational guides
- Health Coaching: Participants in this group received health coaching calls
  Health Coaching Calls: Participants in this group received 12 weekly health coaching calls
Period: Overall Study
Arm/Group | Control Group | Health Coaching
Started | 33 | 30
Completed | 33 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Health Coaching | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age and Sex are unknown for one participant in each arm
  years
    number analyzed (Participants) | 32 | 29 | 61
    (all) | 68.301 (9.562) | 69.410 (6.300) | 68.828 (8.129)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Age and Sex are unknown for one participant in each arm
  Participants
    number analyzed (Participants) | 32 | 29 | 61
    Female | 21 | 16 | 37
    Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 31 | 28 | 59
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 30 | 22 | 52
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Dyspnea Score
Description: The CRQ-Dyspnea is a 5-item questionnaire that assesses dyspnea on a Likert scale from 1 - 7. Higher scores indicate less severity of dyspnea.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Control Group: Participants in this group received 6 educational guides
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 0.29 [-0.02 to 0.59] | -0.26 [-0.66 to 0.14]

2. Primary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Fatigue Score
Description: The CRQ-Fatigue is a 4-item questionnaire that assesses fatigue on a Likert scale from 1 - 7. Higher scores indicate less severity of fatigue.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 0.53 [-0.05 to 1.12] | 0.33 [0.04 to 0.7]

3. Primary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Mastery Score
Description: The CRQ-Mastery is a 4-item questionnaire that assesses mastery on a Likert scale from 1 - 7. Higher scores indicate a higher level of mastering the ability to deal with the symptoms of the disease.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 0.4 [-0.22 to 1.02] | 0.22 [0.12 to 0.56]

4. Primary Outcome: Change in Chronic Respiratory Questionnaire (CRQ) Emotions Score
Description: The CRQ-Emotions is a 7-item questionnaire that assesses emotions on a Likert scale from 1 - 7. Higher scores indicate less severity of emotions.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 0.35 [0.06 to 0.76] | 0.25 [0.06 to 0.55]

5. Secondary Outcome: Change in Daily Physical Activity
Description: Mean change in the number of steps per day
Time Frame: Baseline,3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
steps per day | 174.25 [-794.96 to 1143.46] | -107.88 [-688.47 to 472.72]

6. Secondary Outcome: Change in Self Management
Description: Self-Management Ability Scale-30 item questionnaire measuring ability and function. Total score range is 0-100, higher score indicated better ability and function.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Control Group: Participants in this group received 6 educational guides
  Control: Participants in this group received 6 educational guides and
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 1.78 [-2.89 to 6.45] | -0.7 [-4.42 to 3.02]

7. Secondary Outcome: Change in Meaning in Life Questionnaire (MLQ) - Presence of Meaning
Description: The MLQ is a 10-item questionnaire that assesses quality of life rated on a seven-point scale from 1 = Absolutely Untrue to 7 =Absolutely True. The Presence of Meaning subscale score = subtract the rating for item #9 from 8, then add to the ratings for items 1, 4, 5, and 6. Total Presence of Meaning Scores range between 5 and 35. Higher scores indicate more fullness of meaning a person feels in their life.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | -0.43 [-3.94 to 3.08] | 0.32 [-1.86 to 2.5]

8. Secondary Outcome: Change in Meaning in Life Questionnaire (MLQ) - Search for Meaning
Description: The MLQ is a 10-item questionnaire that assesses quality of life rated on a seven-point scale from 1 = Absolutely Untrue to 7 =Absolutely True. The Search for Meaning subscale score = add together the ratings for items 2, 3, 7, 8, and 10. Total Search for Meaning scores range between 5 and 35. Higher scores indicate more engaged and motivated a person feels to understand and find meaning in their life
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 2.38 [-2.36 to 7.13] | -1.45 [-3.87 to 0.97]

9. Secondary Outcome: Change in Depression
Description: The Patient Health Questionnaire 9-item (PHQ-9) scale used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
Time Frame: Baseline, 3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | -0.57 [-3.19 to 2.05] | 0.13 [-1.97 to 2.24]

10. Secondary Outcome: Change in Anxiety
Description: The General Anxiety Disorder 2-item (GAD 2) scale assess severity of generalized anxiety disorder. Total scores range from 0-6, a higher score indicates greater anxiety.
Time Frame: Baseline,3 months
Population: Data was not collected or analyzed for eight Health coaching subjects and nine Control subjects at 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Health Coaching | Control Group
Number analyzed (Participants) | 22 | 24
score on a scale | 0.27 [-0.63 to 1.17] | 0.05 [-0.7 to 0.79]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 1 year.
Arm/Group | Control Group | Health Coaching
All-Cause Mortality (participants affected / at risk) | 3/33 | 2/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/33 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03837847/Prot_SAP_000.pdf